CLINICAL TRIAL: NCT00797732
Title: Acupuncture for Dysphagia After Chemoradiation Therapy in Head and Neck Cancer Patients: A Pilot Randomized Control Trial
Brief Title: A Pilot Study of Acupuncture Treatment for Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Weidong Lu, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08-169; K01AT004415-01 (NIH); DFCI-08169 (Other: Dana-Farber Cancer Institute)
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Carcinomas, Squamous Cell; Dysphagia
Keywords: acupuncture; dysphagia; chemoradiation related effects; squamous cell carcinoma of the head and neck; nasopharyngeal cancer; oropharynx cancer; hypopharynx cancer; larynx cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Deglutition Disorders; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Acupuncture (Active Comparator): The active intervention used a three-phase step-up protocol to gradually increase the body areas treated and needling intensity. Acupuncture needles (0.20x25mm) were inserted with a depth of 5-10 mm into predefined points based on a systematic literature review following the STRICTA guideline. Needles were stimulated to obtain the de qi sensation. An electroacupuncture (EA) device was connected at two acupoints. All needles remained in place for 30 minutes. The active acupuncture was administered once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT. [Refs: Lu W, Wayne PM et al. Contemp Clin Trials 2012; 33; 700-711; MacPherson H, Altman DG et al. PLoS Med 2010;7:e1000261]
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): The sham intervention was designed to be maximally inert and minimally invasive, while simulating most aspects of the active protocol. Sham needles (0.12x30mm) were inserted at 14 locations paralleling the same body regions needled in the active group; however, all sham point locations were off the pathways of traditional Chinese medicine acupuncture meridians and points. An identical but deactivated EA device was used following sham protocols previously used. The sham acupuncture was administered once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT. [Refs: Lu W, Wayne PM et al. Contemp Clin Trials 2012; 33; 700-711; Wayne PA, Krebs DE et al. Arch Phys Med Rehabil 2005;86:2248-2255]
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
The current standard of care for advanced HNC is concurrent chemoradiation therapy (CRT), which has led to increased survival rates, but with significant acute and long-term toxicities. Dysphagia, or difficulty with swallowing, is a common and expected side effect during and following CRT. Dysphagia occurs in up to 50% of patients and significantly impairs the quality of life (QOL) of patients during delivery of and recovery from CRT. Clinical trials evaluating promising and innovative adjunctive approaches that could increase the rate and magnitude of recovery from dysphagia in HNC patients are needed. Acupuncture is a traditional Chinese medical technique that has been found to reduce symptoms and side effects associated with primary cancer therapy. This study evaluated the feasibility of conducting a randomized sham-controlled trial and collected preliminary data on safety and efficacy of acupuncture.

DETAILED DESCRIPTION:
AIMS:

Aim 1. To assess the feasibility of recruiting and retaining HNC patients with dysphagia into a randomized sham-controlled trial of acupuncture.

Aim 2. To collect preliminary data on the efficacy of acupuncture in changing scores of HRQOL in post CRT head and neck cancer patients.

Aim 3. (Exploratory) In a subset of HNC subjects treated with both active and sham acupuncture, to collect objective measures on swallowing functions using Videofluoroscopic swallowing study (VFSS); salivary flow production; and plasma Transforming Growth Factor (TGF)-β1, Interleukin 6 (IL-6), Tumor necrosis factor-alpha (TNF-α) and Interleukin 13 levels.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck (SCCHN) at stage II, III and IV, without evidence of distant metastasis. Stage I disease will also be permitted if the patient is receiving CRT;
* Primary tumor sites eligible: nasopharyngeal, oropharynx, hypopharynx or larynx. Tumors of the nasal and paranasal cavities will also be included. Unknown primary squamous cell carcinoma (SCC) in the neck will also be eligible. SCC of the oral cavity will also be eligible with the approval of the treating staff;
* Receiving chemoradiation;
* Currently or recently undergoing swallowing therapy program with or without feeding tube use, with or without neck dissection;
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Adequate hematological function: neutrophil count >1.0 x109/L, platelet count >50x109/L
* Signed informed consent.

Exclusion Criteria

Patients with the following criteria will NOT be eligible for the study:

* Unstable cardiac disease or myocardial infarction within 6 months prior to study entry;
* Wearing a pacemaker or implantable cardioverter-defibrillator;
* History of significant neurologic disorder that affects swallowing, including stroke, neurodegenerative disease, advanced dementia, or uncontrolled seizure disorder;
* Active clinically significant uncontrolled infection;
* Prior use of acupuncture for dysphagia;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-12; Primary Completion 2013-01 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Lu, MB, MPH, PhD, Principal Investigator — Harvard Medical School/Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu W, Wayne PM, Davis RB, Buring JE, Li H, Goguen LA, Rosenthal DS, Tishler RB, Posner MR, Haddad RI. Acupuncture for dysphagia after chemoradiation in head and neck cancer: rationale and design of a randomized, sham-controlled trial. Contemp Clin Trials. 2012 Jul;33(4):700-11. doi: 10.1016/j.cct.2012.02.017. Epub 2012 Mar 2. PMID 22406102
- [Background] Lu W, Posner MR, Wayne P, Rosenthal DS, Haddad RI. Acupuncture for dysphagia after chemoradiation therapy in head and neck cancer: a case series report. Integr Cancer Ther. 2010 Sep;9(3):284-90. doi: 10.1177/1534735410378856. Epub 2010 Aug 16. PMID 20713374
- [Background] Lu W, Wayne PM, Davis RB, Buring JE, Li H, Macklin EA, Lorch JH, Burke E, Haddad TC, Goguen LA, Rosenthal DS, Tishler RB, Posner MR, Haddad RI. Acupuncture for Chemoradiation Therapy-Related Dysphagia in Head and Neck Cancer: A Pilot Randomized Sham-Controlled Trial. Oncologist. 2016 Dec;21(12):1522-1529. doi: 10.1634/theoncologist.2015-0538. Epub 2016 Aug 10. PMID 27511906
- [Derived] Lu W, Giobbie-Hurder A, Tanasijevic A, Baedorf Kassis S, Park SH, Jeong YJ, Shin IH, Yao C, Jung HJ, Zhu Z, Bao C, Yang EM, Bierer BE, Ligibel JA. Acupuncture for hot flashes in hormone receptor-positive breast cancer, a coordinated multinational study: Rationale and design of the study protocol. Contemp Clin Trials. 2022 Oct;121:106885. doi: 10.1016/j.cct.2022.106885. Epub 2022 Aug 20. PMID 35998768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for potential enrollment from January 2009 through December 2011.
Pre-assignment Details: Since one primary aim was to assess feasibility as measured by recruitment the screening non-randomized count is included in the participant flow.
Groups:
- Sham Acupuncture: The sham intervention was designed to be maximally inert and minimally invasive, while simulating most aspects of the active protocol. Sham needles (0.12x30mm) were inserted at 14 locations paralleling the same body regions needled in the active group; however, all sham point locations were off the pathways of traditional Chinese medicine acupuncture meridians and points. An identical but deactivated EA device was used following sham protocols previously used. The sham acupuncture was administered once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT. [Refs: Lu W, Wayne PM et al. Contemp Clin Trials 2012; 33; 700-711; Wayne PA, Krebs DE et al. Arch Phys Med Rehabil 2005; 86:2248-2255]
- Screened Non-Randomized: Participants approached in the screening process but ultimately not randomized.
Period: Overall Study
Arm/Group | Active Acupuncture | Sham Acupuncture | Screened Non-Randomized
Started | 21 | 21 | 154
Evaluable at Baseline (Evaluable for quality of life assessment.) | 18 | 18 | 0
Evaluable at 20 Weeks (Evaluable for quality of life assessment.) | 17 | 18 | 0
Evaluable at 12 Months (Evaluable for quality of life assessment.) | 17 | 18 | 0
Completed | 16 | 18 | 0
Not Completed | 5 | 3 | 154
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Not meet inclusion criteria | 0 | 0 | 7
Not completed — Excluded due to time constraints | 0 | 0 | 24
Not completed — Refused to Participate | 0 | 0 | 123

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all randomized participants.
Groups:
- Active Acupuncture: Both active and sham acupuncture were administered by 5 experienced staff acupuncturists employing a traditional Chinese medicine (TCM) style, once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT.
- Sham Acupuncture: TBoth active and sham acupuncture were administered by 5 experienced staff acupuncturists employing a traditional Chinese medicine (TCM) style, once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT.
- Total: Total of all reporting groups
Arm/Group | Active Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.8) | 59.1 (8.3) | 58.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 18 | 16 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42
Total IMRT dose (Gy) [Count of Participants; unit: Participants] — IMRT, intensity modulated radiation therapy, dose received
  Participants
    58 Gy | 1 | 0 | 1
    64 GY | 0 | 3 | 3
    66 Gy | 1 | 2 | 3
    70 Gy | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Outcome Compliance Rate
Description: Outcome compliance rate is the percentage of enrolled participants who completed the primary study assessments (at baseline and in long-term follow-up 6 months post acupuncture treatment).
Time Frame: Assessed at baseline and at 6 months post acupuncture treatment
Population: The analysis population is comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Sham Acupuncture: Both active and sham acupuncture were administered by 5 experienced staff acupuncturists employing a traditional Chinese medicine (TCM) style, once every 2 weeks for 24 weeks, starting 2 weeks into CRT and ending at 20 weeks after CRT.
Arm/Group | Active Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 21 | 21
percentage of participants | 76.2 [52.8 to 91.8] | 85.7 [63.6 to 97.0]

2. Primary Outcome: Treatment Compliance Rate
Description: Treatment compliance rate is the percentage of enrolled participants who completed at least 80% of treatment (10 of 12 acupuncture sessions).
Time Frame: Assessed throughout the 6 month treatment period (12 acupuncture treatments every 2 weeks)
Population: The analysis population is comprised of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 21 | 21
percentage of participants | 76.2 [52.8 to 91.8] | 81.0 [58.1 to 94.6]

3. Secondary Outcome: MDADI Change From Baseline to 12 Months Post Chemoradiation Therapy (CRT)
Description: The M.D. Anderson Dysphagia Inventory (MDADI) is a validated, self-administered questionnaire established as the best measure of dysphagia-related quality of life in HNC patients. (Carlsson S, et al Dysphagia 2012; 27: 361-369). MDADI has two summary scores: 1) global (1 item) and 2) composite (19 items). Each item is scored on a 5 point Likert scale (strongly disagree, disagree, no opinion, agree, strongly agree). The composite MDADI score is a weighted average of the physical, emotional, and functional subscale questions. Scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning). A minimal clinically important within group difference was a 10% change from baseline.
Time Frame: Assessed at baseline and 6 months post acupuncture which parallels 12 months post-CRT
Population: The analysis population represents the subset of participants evaluable at baseline and 12 months post CRT/6 months post acupuncture
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 16 | 18
units on a scale | 7.9 [0.2 to 15.6] | 13.9 [6.4 to 21.4]
Statistical Analysis 1: Comparison: Active Acupuncture vs Sham Acupuncture; Test type: Superiority; p = .17, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: MDADI Scores
Description: as for outcome 3
Time Frame: Assessed at baseline, 20 weeks post chemoradiation therapy and 6 months post acupuncture
Population: The analysis population is comprised of all randomized participants. At each timepoint, a subset of participants were evaluable for quality of life assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline: number analyzed (Participants) | 18 | 18
  Baseline | 60.3 (14.7) | 69.2 (15.5)
  20 weeks post chemoradiation start: number analyzed (Participants) | 17 | 18
  20 weeks post chemoradiation start | 68.7 (13.3) | 77.8 (10.9)
  6 months post acupuncture start: number analyzed (Participants) | 16 | 18
  6 months post acupuncture start | 72.7 (13.3) | 79.3 (12.4)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated throughout treatment at each visit up to end of treatment week 20 after CRT.
Arm/Group | Active Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Acupuncture (N=21) | Sham Acupuncture (N=21)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No